CLINICAL TRIAL: NCT02443597
Title: Can Increased Body Mass Index Prevent Adequate Ultrasound Examination for Trisomy 21 Risk Assessment?
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Collaborators: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, ahmed abdulmoneim altraigey, lecturer, Benha University
Other Study IDs: AFHSRMREC/2015/OB/GYNAE/053
Record Dates: First submitted 2015-05-02; First posted 2015-05-14 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Ultrasound Quality
Keywords: ultrasound; trisomy screening; obesity
MeSH Terms: conditions — Obesity | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- obese pregnant women: With the use of trans-abdominal ultrasound, the following measurements will be recorded:
  * Fetal nuchal translucency thickness.
  * Nasal bone.
  * Fetal facio-maxillary angle.
  * The flow across the tricuspid valve as normal or regurgitated.
  * A-wave in the ductus venosus as normal or reversed.
  Interventions: Other: ultrasound
- lean pregnant women: With the use of trans-abdominal ultrasound, the following measurements will be recorded:
  * Fetal nuchal translucency thickness.
  * Nasal bone.
  * Fetal facio-maxillary angle.
  * The flow across the tricuspid valve as normal or regurgitated.
  * A-wave in the ductus venosus as normal or reversed.
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — trans abdominal or trans vaginal ultrasound to detect some of the soft markers of trisomy screening

SUMMARY:
Determine Cutoff BMI at which transabdominal sonography (TAS) is not satisfactory for aneuploidy risk assessment.

DETAILED DESCRIPTION:
Obesity is a common public health problem which is increasing worldwide at an alarming rate. According to National nutrition survey statistics of 2007, the prevalence of obesity in the kingdom of Saudi Arabia was 23.6% in women and 14% in men. Also the prevalence of overweight in the Saudi community was determined to be 30.7% for men as compared to 28.4% for the women.

First trimester screening between 11-14 weeks gestation is known to be an effective and reliable screening test for Down syndrome and trisomy 18.First trimester screening allows earlier identification of the pregnancy at risk for fetal aneuploidy and anatomic defects, particularly, cardiac anomalies, therefore, providing an option of earlier diagnosis by chorionic villus sampling and analysis of amniocytes.

The well-known association of obesity during pregnancy with a variety of maternal and fetal complications increases the importance of early aneuploidy screening.

Fetal aneuploidy risk assessment is based on a combination of maternal age, prior affected pregnancy or family history, maternal serum biochemical tests and fetal ultrasound markers.

The impact of obesity on the quality of prenatal ultrasound examination is well established with a greater risk for suboptimal visualization, in particular, the fetal cardiac structures and the craniospinal structures only when body mass index above the 90th percentile.

The quality of prenatal screening for aneuploidy via nuchal translucency thickness measurement is significantly limited among obese pregnant women, thus, increased risk of fetal anomalies.

Gandhiet al, have noted that increased BMI is not associated with suboptimal visualization of nuchal translucency, but it is associated with a longer time to perform the first-trimester ultrasound examination for aneuploidy risk assessment, increased need for transvaginal ultrasound examination for optimum nuchal translucency visualization.

There is evidence suggesting that fetal anatomic evaluation in the low-risk gravida can be better accomplished in the first trimester using the transvaginal route, providing a valuable option for obese patients.

ELIGIBILITY:
Inclusion Criteria:

* women who have a live, intrauterine, singleton pregnancy between 11- 14 weeks gestation.

Exclusion Criteria:

* multiple gestation.
* fetal size outside of nuchal translucency screening age (crown-rump length (CRL) outside of 46-71 mm).
* presence of a cystic hygroma.
* fetal demise.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Inclusion criteria will consist of women who have a live, intrauterine, singleton pregnancy between 11- 14 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Cutoff body mass index for the use of transvaginal ultrasound for aneuploidy risk assessment. | 30 minutes

SECONDARY OUTCOMES:
The time of the study. (time needed for satisfactory ultrasound risk assessment in minutes) | 30 minutes
  time needed for satisfactory ultrasound risk assessment in minutes
The tolerance of the woman for trans-vaginal ultrasound. | 30 minutes
  preference of the patients towards transabdominal and transvaginal ultrasound
The harmful effect to the patient | 12 hours
  Infection, Bleeding, Injury to vagina or cervix and uterine irritability.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed altraigey, Study Director — Benha University; haytham atia, Principal Investigator — Zagazig University; nuzhat amer, Principal Investigator — Armed Forces Hospitals, Southern Region, Saudi Arabia; Mohamed Kolkailah, Study Chair — Armed Forces Hospitals, Southern Region, Saudi Arabia; mohammed ellaithy, Principal Investigator — Ain Shams University; magdy eldumairy, Principal Investigator — Armed Forces Hospitals, Southern Region, Saudi Arabia
Locations (1):
- antenatal clinic of Armed Forces Hospital, Southern Region, Khamis Mushait, 'Asir Region, Saudi Arabia